CLINICAL TRIAL: NCT06196892
Title: A Randomized, Double-blind Controlled Trial to Assess the Impact of Probiotic on the Intestinal Health of Individuals
Brief Title: Probiotics Improve Health Young Volunteers' Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023007
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): one sachet per day, with maltodextrin
  Interventions: Dietary Supplement: Placebo
- Probiotic group (Experimental): one sachet per day, with BBr60 and maltodextrin
  Interventions: Dietary Supplement: Probiotic BBr60

INTERVENTIONS:
Dietary Supplement: Probiotic BBr60 — Collect patient fecal samples, test for 16S rRNA, and analyze the changes in the patient's gut microbiota before and after taking BBr60.
  Arms: Probiotic group
Dietary Supplement: Placebo — Collect patient fecal samples, test for 16S rRNA, and analyze the changes in the patient's gut microbiota before and after taking maltodextrin.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate whether daily supplementation with the probiotic Bifidobacterium breve BBr60 can improve metabolic, gastrointestinal, and emotional health in healthy adult volunteers aged 19 to 45 years.

The main questions it aims to answer are: Can B. breve BBr60 improve lipid metabolism (e.g., increase HDL and reduce total cholesterol) in healthy adults? Can B. breve BBr60 alleviate gastrointestinal symptoms and improve emotional well-being in a non-clinical population? Researchers will compare a BBr60 supplementation group to a placebo group to see if the probiotic group experiences greater improvements in metabolic, gastrointestinal, and psychological indicators.

Participants will: Take one sachet daily of either B. breve BBr60 (10 billion CFU) or placebo for 8 weeks. Provide blood and stool samples at baseline and week 8. Complete validated questionnaires assessing alcohol dependence, gastrointestinal symptoms, and emotional status.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19-45 years;
2. Willing to voluntarily agree to and comply with the trial protocol, and capable of timely participation in screening and follow-up;
3. Have not suffered from gastrointestinal diseases in the past month;
4. Have not taken antibiotics in the past month.

Exclusion Criteria:

1. Individuals under 19 or over 45 years of age, with an allergic constitution or allergy to any component of the test substance, symptoms of alcohol allergy, and pregnant or breastfeeding women;
2. Those who experience discomfort such as diarrhea or bloating after taking the test substance;
3. Patients with serious diseases of the cardiovascular, liver, kidney, hematopoietic systems, autoimmune diseases, endocrine disorders, mental illnesses, existing high blood sugar, or unhealthy gastrointestinal conditions;
4. Those who discontinue the test sample or take other medications midway, making it difficult to judge efficacy or with incomplete data;
5. Recently taken probiotics, prebiotics, or antibiotics related to the function of the test substance, affecting the judgment of results;
6. Individuals with a daily diet that is either too light or too greasy; those with special dietary structures due to weight loss or other reasons (such as a ketogenic diet);
7. Individuals with low body fat, BMI < 23.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Changes in intestinal flora | 8 weeks
  Collect patient fecal samples, test for 16S rRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Kang Zou, Nanjing, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong Y, Cai Y, Tian H, Wen J, Han M, Tan Y, Zou K. The impact of Bifidobacterium breve BBr60 (BBr60) on metabolic and gastrointestinal health in healthy adults: A combined in vitro metabolomic and randomized, double-blind, placebo-controlled study. Clin Nutr. 2025 Aug;51:349-361. doi: 10.1016/j.clnu.2025.07.004. Epub 2025 Jul 7. PMID 40652782